CLINICAL TRIAL: NCT02158299
Title: Contrast The Role of Microfibrillar Collagen Hemostat Flour（Avitene） And OK-432 （Sapylin）in Reducing Seroma Formation After Axillary Lymphadenectomy for Breast Cancer
Brief Title: Contrast The Role of Avitene And OK-432 in Reducing Seroma Formation After Axillary Lymphadenectomy for Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Jia Weijuan, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Clinical trail003
Record Dates: First submitted 2014-05-22; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Drainage; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Collagen; streptococcal preparation 722

STUDY DESIGN:
Who Masked: Care Provider

ARMS (3):
- Avitene,Drainaging,reexamine (Experimental)
  Interventions: Drug: Avitene; Behavioral: axillary drainage; Other: reexamine
- Sapylin,Drainaging,reexamine (Experimental)
  Interventions: Drug: Sapylin; Behavioral: axillary drainage; Other: reexamine
- Drainaging,reexamine (Active Comparator)
  Interventions: Behavioral: axillary drainage; Other: reexamine

INTERVENTIONS:
Drug: Avitene
  Arms: Avitene,Drainaging,reexamine
Drug: Sapylin
  Arms: Sapylin,Drainaging,reexamine
Behavioral: axillary drainage
Other: reexamine

SUMMARY:
After Axillary lymphadenectomy for breast cancer there are not few patients showed seroma formation and it can not be ignored.Investigators aimed to study two new methods of application of Microfibrillar Collagen Hemostat Flour and OK-432 to reduce seroma formation and to verify the efficacy and safety of these two applications.Try to prove them as beneficial supplements for axillary lymphadenectomy of breast cancer.

DETAILED DESCRIPTION:
A prospective,randomized analysis of breast-conserving surgery or mastectomy plus axillary lymphadenectomy for those patients with sentinel node positive using Microfibrillar Collagen Hemostat Flour 、 OK-432 or using nothing in equal probability.Up to 12 months,a total of 180 will be recruited in plan.During the operation and after the axillary lymphadenectomy，according the arms，Investigators put Microfibrillar Collagen Hemostat Flour（avitene）、 OK-432（Sapylin） or nothing into patients axillary wounds。And Investigators will the statistical significance of these three arms that the postoperative drainage magnitude and duration.Also the complications associated with axillary lymphadenectomy will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered for the study and signed informed consent；
2. Preoperative biopsy or intraoperative sentinel lymph node biopsy confirmed axillary lymph node metastasis and need axillary lymphadenectomy
3. No penicillin allergy
4. No blood system diseases
5. No rheumatic heart disease
6. No history or family history of asthma
7. No history of axillary surgery

Exclusion Criteria:

1. A history of severe hypertension
2. A history of diabetes
3. Undergoing anticoagulant therapy or anticoagulant therapy drug withdrawal less than a year
4. BMI>30
5. Can not accept telephone follow-up or can not go to the hospital for subsequent inspection treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
postoperative drainage magnitude | up to 1 year

SECONDARY OUTCOMES:
Duration of the drainage | up to 1 year

OTHER OUTCOMES:
The complications of seroma formation | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jia Wei juan, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China